CLINICAL TRIAL: NCT04904575
Title: Erector Spinae Plane Block in Lumbar Spinal Fusion : Double-blind, Randomized Controlled Trial.
Brief Title: Erector Spinae Plane Block in Lumbar Spinal Fusion
Acronym: MERFUSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL2020-GL01
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spinal Fusion
Keywords: Erector spinae plane block; consumption of morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block (Experimental): The "Block" group will be made up of patients who will benefit from an injection of levobupivacaine for the realization of the erector spinae plane block.
  Interventions: Procedure: Erector spinae plane block
- Placebo (Placebo Comparator): The "placebo" group corresponds to the reference group, that is to say that it will consist of patients who will benefit from an injection of physiological serum for the realization of the erector spinae plane block.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Procedure : After installing the sleeping patient and identifying the surgical level by the surgeon, the anesthetist will perform the erector spinae plane block. The anesthetist performs an ultrasound to view the spine and erector muscles and identifies the transverse processes of the vertebra involved in the surgery. Once the location has been made, the anesthetist injects the anesthetic product under ultrasound control between the erector muscle of the spine and its anterior fascia, the trajectory of the needle being thus visualized throughout the procedure. The anesthetist bilaterally injects 3ml/kg of solution with a maximum of 30ml injected.
  Drug : Levobupivacaïne 2,5mg/ml.
  Arms: Block
Procedure: Erector spinae plane block — Procedure : After installing the sleeping patient and identifying the surgical level by the surgeon, the anesthetist will perform the erector spinae plane block. The anesthetist performs an ultrasound to view the spine and erector muscles and identifies the transverse processes of the vertebra involved in the surgery. Once the location has been made, the anesthetist injects the anesthetic product under ultrasound control between the erector muscle of the spine and its anterior fascia, the trajectory of the needle being thus visualized throughout the procedure. The anesthetist bilaterally injects 3ml/kg of solution with a maximum of 30ml injected.
  Drug : NaCL 0,9%.
  Arms: Placebo

SUMMARY:
The aim of this study is to observe or not a reduction in the consumption of morphine within 72 hours of the realization of an erector spinae plane block when preparing for a lumbar spinal fusion.

DETAILED DESCRIPTION:
Posterior lumbar spine surgery is surgery described by patients as painful. For this type of surgery, lumbar spinal fusion, especially because of greater exposure, is more painful than simple surgeries to release the lumbar canal or to cure a herniated disc. However, the improvement of implants and techniques, as well as the change in the habits of surgeons, means that this lumbar spinal is on the increase (+ 65%). The management of postoperative pain is a priority for anesthesiologic teams with a goal to improved rehabilitation after surgery.

Multimodal analgesia, already recognized for other surgeries, is one of the keys to success, combining oral analgesics and regional local anesthetics.

The recourse to the realization of a erector spinae plane block was described for the first time in 2016, it is described as not presenting any particular risk, simple to apply and having a satisfactory analgesia action. However, this process is little described in the context of spine surgery and even less in the context of randomized controlled trials. On the other hand, no study has evaluated the effectiveness of spinal block as part of an Enhanced Rehabilitation After Surgery (RAAC) program.

At the Clinique Saint Jean Sud de France, the management of spine surgeries is part of an Improved Rehabilitation After Surgery (RAAC) process. Patients benefit from multidisciplinary preoperative information and perioperative management promoting early mobilization and postoperative rehabilitation.

It seemed relevant to carry out a randomized, controlled, double-blind study to evaluate the consumption of postoperative morphine during the 72 hours following a lumbar spinal fusion.

The studied process will be the realization of a ultrasound guided erector spinae plane block.

The realization of the erector spinae plane block is carried out as part of lumbar spinal fusion surgery on 1 or 2 levels.

As part of this study, 130 patients will be randomized into 2 arms: one arm receiving the anesthetic and another arm receiving the placebo. As the study is double blind, both arms will benefit from the same procedure. Patients in the block arm will receive an injection of levobupivacaine 2.5 mg / ml while the patients in the placebo arm will receive an injection of physiological saline (NaCL 0,9%) in the same proportions.

The data necessary for this study will be collected directly from the patient and from his medical file according to the following schedule: 3h, 4h, 6h, 9h, 12h, 18h, 24h, 36h, 48h, 72h and 1 month after realization of the erector spinae plane block.

ELIGIBILITY:
Inclusion Criteria:

* Patient with medical insurance.
* Patient who received information about study and signes a consent to participate in the study.
* Major patient requiring a lumbar spinal fusion surgery.
* Patient with an ASA score of 1, 2 or 3.

Exclusion Criteria:

* Minor patient.
* Patient with morphine intolerance
* Patient with allergy to local anesthetics.
* Patient consuming morphine for more than 3 months.
* Pregnant or breastfeeding patient.
* Patient scheduled for cancer surgery or trauma surgery.
* Patient participating in another interventional study.
* Patient with history of lumbar spinal fusion.
* Patient requiring lumbar surgery without arthrodesis.
* Patient requiring lumbar surgery with inter-lamar or inter-epineal stabilization.
* Patient refusing to sign the consent form.
* Patient for whom it is impossible to give informed information.
* Patient under the protection of justice, under curatorship or under tutorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Consumption of postoperative morphine within 72 hours of the operation. | 72 hours

SECONDARY OUTCOMES:
Digital visual scale to assess pain of patient within 72 hours of the operation. | 72 hours
  Numeric scale numbered from 0 to 10. 0 : no pain, 10: worst pain possible
Onset of nausea and vomiting within 72 hours of the operation. | 72 hours
  Onset of nausea/ vomiting or taking an anti-vomiting treatment within 72 hours of the operation.
Onset of complication within 30 days of the intervention. | 30 days
Walking perimeter measurement by the physiotherapist during the 72 hours following the intervention. | 72 hours
  Measurement of the maximum distance traveled without stopping in meter with or without assistance.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LONJON, MD, Principal Investigator — Clinique Saint Jean, Saint Jean de Védas
Locations (1):
- Clinique Saint Jean, Saint-Jean-de-Védas, France

REFERENCES:
- [Background] Chen K, Wang L, Ning M, Dou L, Li W, Li Y. Evaluation of ultrasound-guided lateral thoracolumbar interfascial plane block for postoperative analgesia in lumbar spine fusion surgery: a prospective, randomized, and controlled clinical trial. PeerJ. 2019 Oct 28;7:e7967. doi: 10.7717/peerj.7967. eCollection 2019. PMID 31681518
- [Background] Ren Z, Li Z, Li S, Sheng L, Xu D, Chen X, Wu WKK, Chan MTV, Ho J. Local infiltration with cocktail analgesics during 2 level lumbar spinal fusion surgery: Study protocol of a randomized controlled trial. Medicine (Baltimore). 2019 May;98(19):e15526. doi: 10.1097/MD.0000000000015526. PMID 31083198
- [Background] Breebaart MB, Van Aken D, De Fre O, Sermeus L, Kamerling N, de Jong L, Michielsen J, Roelant E, Saldien V, Versyck B. A prospective randomized double-blind trial of the efficacy of a bilateral lumbar erector spinae block on the 24h morphine consumption after posterior lumbar inter-body fusion surgery. Trials. 2019 Jul 17;20(1):441. doi: 10.1186/s13063-019-3541-y. PMID 31315670
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Qiu Y, Zhang TJ, Hua Z. Erector Spinae Plane Block for Lumbar Spinal Surgery: A Systematic Review. J Pain Res. 2020 Jul 1;13:1611-1619. doi: 10.2147/JPR.S256205. eCollection 2020. PMID 32669870
- [Background] Ince I, Atalay C, Ozmen O, Ozturk V, Hassan M, Aksoy M, Calikoglu C. Comparison of ultrasound-guided thoracolumbar interfascial plane block versus wound infiltration for postoperative analgesia after single-level discectomy. J Clin Anesth. 2019 Sep;56:113-114. doi: 10.1016/j.jclinane.2019.01.017. Epub 2019 Feb 8. No abstract available. PMID 30743153
- [Background] Cesur S, Yayik AM, Ozturk F, Ahiskalioglu A. Ultrasound-guided Low Thoracic Erector Spinae Plane Block for Effective Postoperative Analgesia after Lumbar Surgery: Report of Five Cases. Cureus. 2018 Nov 16;10(11):e3603. doi: 10.7759/cureus.3603. PMID 30680264
- [Background] Mathiesen O, Dahl B, Thomsen BA, Kitter B, Sonne N, Dahl JB, Kehlet H. A comprehensive multimodal pain treatment reduces opioid consumption after multilevel spine surgery. Eur Spine J. 2013 Sep;22(9):2089-96. doi: 10.1007/s00586-013-2826-1. Epub 2013 May 17. PMID 23681498
- [Background] Davies AF, Segar EP, Murdoch J, Wright DE, Wilson IH. Epidural infusion or combined femoral and sciatic nerve blocks as perioperative analgesia for knee arthroplasty. Br J Anaesth. 2004 Sep;93(3):368-74. doi: 10.1093/bja/aeh224. Epub 2004 Jul 9. PMID 15247111
- [Background] Benyahia NM, Verster A, Saldien V, Breebaart M, Sermeus L, Vercauteren M. Regional anaesthesia and postoperative analgesia techniques for spine surgery - a review. Rom J Anaesth Intensive Care. 2015 Apr;22(1):25-33. PMID 28913452
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Kendall MC, Alves L, Traill LL, De Oliveira GS. The effect of ultrasound-guided erector spinae plane block on postsurgical pain: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 May 1;20(1):99. doi: 10.1186/s12871-020-01016-8. PMID 32357842
- [Background] Nielsen RV, Fomsgaard JS, Dahl JB, Mathiesen O. Insufficient pain management after spine surgery. Dan Med J. 2014 May;61(5):A4835. PMID 24814741
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233